CLINICAL TRIAL: NCT04744194
Title: The Effect of a 6 Week Nordic Hamstring Exercise and an Assisted Nordic Hamstring Program on Hamstring Muscle Strength
Brief Title: The Effect of 6 Week Hamstring Exercise Programs on Hamstring Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dublin City University (Other)
Responsible Party: Principal Investigator, Enda Whyte, Assistant Professor, Dublin City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019_10_EW/FB
Record Dates: First submitted 2021-02-01; First posted 2021-02-08 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Hamstring Injury
Keywords: Eccentric hamstring strength; Nordic hamstring exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic hamstring exercise program (Active Comparator): Participants are required to kneel on a gym mat keeping their hips in a slightly flexed position and to slowly lower themselves in a controlled manner as far as they could towards the ground. When they can no longer lower themselves as such, they are instructed to utilise their arms to buffer the fall and touch their chest off the ground, while maintaining tension in their hamstrings. Once their chest touches the ground they are instructed to immediately return to the starting position by pushing up with their hands
  Interventions: Other: Nordic hamstring exercise program
- Assisted nordic hamstring exercise program (Experimental): Participants are required to kneel on a gym mat keeping their hips in a slightly flexed position and to slowly lower themselves in a controlled manner as far as they could towards the ground. During this exercise, participants are attached to a weighted pulley cable system via a chest attachment. A sufficient amount of assistance is given to allow the participant to lower to 30 degrees of knee flexion. When they can no longer lower themselves as such, they are instructed to utilise their arms to buffer the fall and touch their chest off the ground, while maintaining tension in their hamstrings. Once their chest touches the ground they are instructed to immediately return to the starting position by pushing up with their hands
  Interventions: Other: Assisted nordic hamstring exercise program

INTERVENTIONS:
Other: Nordic hamstring exercise program — Week 1 - 1 session per week consisting of 2 sets of 5 reps of the exercise Week 2 - 2 sessions per week consisting of 2 sets of 6 reps of the exercise Week 3 - 3 sessions per week consisting of 3 sets of 6 reps of the exercise Week 4 - 3 sessions per week consisting of 3 sets of 8 reps of the exercise Weeks 5 and 6 - 3 sessions per week consisting of 3 sets of the exercise. Set 1 with 12 reps, set 2 with 10 reps and set 3 with 8 reps.
  Arms: Nordic hamstring exercise program
Other: Assisted nordic hamstring exercise program — Week 1 - 1 session per week consisting of 2 sets of 5 reps of the exercise Week 2 - 2 sessions per week consisting of 2 sets of 6 reps of the exercise Week 3 - 3 sessions per week consisting of 3 sets of 6 reps of the exercise Week 4 - 3 sessions per week consisting of 3 sets of 8 reps of the exercise Weeks 5 and 6 - 3 sessions per week consisting of 3 sets of the exercise. Set 1 with 12 reps, set 2 with 10 reps and set 3 with 8 reps.
  Arms: Assisted nordic hamstring exercise program

SUMMARY:
This study aims to compare the effect of two hamstring strengthening programs on hamstring muscle strength in university students. 60 participants will be recruited for this study. They will be randomly assigned to one of two 6-week hamstring strengthening programs, namely the single leg bridge exercise and the Nordic hamstring exercise protocol, and one control group. Eccentric and isometric hamstring strength, gluteal strength and will sprint speed will be measured before and after the intervention.

DETAILED DESCRIPTION:
Participants will be recruited from the local university sports clubs. Club chairpersons will be asked to send an email to club players. Players interested in participating in the study will be asked to attend a meeting where the study will be explained to them. Those who were interested will then be assessed for inclusion and exclusion criteria.

Group allocation:

A four block randomization method will be used to allocate participants to the Nordic hamstring exercise protocol or the single leg bridge protocol.

Interventions:

The Nordic hamstring exercise program or the single leg bridge program.

Testing procedure:

The eccentric strength of the participants' hamstrings will be recorded before and after the exercise intervention.

A 10 point visual analogue scale will be used to record the level of muscle soreness experienced after each training session.

ELIGIBILITY:
Inclusion Criteria:

* free from hamstring injury in the 6 months prior to the study
* currently competing in team sports at least three occasions per week

Exclusion Criteria:

* history of a hip or knee injury in the 3 months prior to the study
* a history of anterior cruciate ligament rupture
* a history of involvement in a hamstring strengthening, injury prevention programme in the 3 months prior to the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-02-13 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
Eccentric hamstring strength | Change from baseline after 6 weeks
  This will be measured using devices that measure the eccentric strength of the hamstrings during the Nordic hamstring exercise. The devices are called the Hamstring Solo device and the Nordbord device. Participants will kneel on the padded surface of the device with their lower limbs held in position just above the ankles. The ankle supports have load sensitive cells. The participants will be asked to complete the nordic hamstring exercise. This involves them folding their arms across their chest and slowly lowering themselves towards the ground by allowing their knees to slowly straighten. The load cells will record the force (newtons) during the exercise for each leg.
Eccentric hamstring moment | Change from baseline after 6 weeks
  This will be measured using devices that measure the eccentric strength of the hamstrings during the Nordic hamstring exercise. The devices are called the Hamstring Solo device and the Nordbord device. Participants will kneel on the padded surface of the device with their lower limbs held in position just above the ankles. The ankle supports have load sensitive cells. The participants will be asked to complete the nordic hamstring exercise. This involves them folding their arms across their chest and slowly lowering themselves towards the ground by allowing their knees to slowly straighten. The load cells will record the force (newtons) during the exercise for each leg. The distance from the load cells to the knee joint will be measured (meters) to calculate the moment in Newton meters for the exercise
Hamstring strength endurance | Change from baseline after 6 weeks
  This will be measured by assessing the number of repetitions of the single leg bridge exercise to failure

SECONDARY OUTCOMES:
Muscle soreness ratings following exercise | immediately following each session
  Participants will use a ten point numerical rating scale to record the level of muscle soreness after training sessions. The scale will range from 0 to 10 where 0 is no pain and 10 is the most severe pain imaginable.
between limb asymmetries in hamstring strength, moment and endurance. | Change from baseline after 6 weeks
  percentage between limb asymmetries will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: enda whyte, PhD, Principal Investigator — Dublin City University
Locations (1):
- Dublin City University, Dublin, Ireland